CLINICAL TRIAL: NCT06258889
Title: Optimizing Exposure Therapy Via Reward-focused Interventions: A Randomized Controlled Trial in Individuals With Public Speaking Anxiety
Brief Title: Optimizing Exposure Therapy Via Reward-focused Interventions in Individuals With Public Speaking Anxiety
Acronym: EXOPAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Christoph Benke, Principal Investigator, Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EXOPAT_SPEAKING_ANX
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Public Speaking Fear
MeSH Terms: conditions — Glossophobia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- reward-focused intervention + exposure (Experimental): Psychoeducation reward-focused interventions based on Positive Affect Treatment (Finding the silver lining, taking ownership, imagining the positive) Exposure & reward-focused interventions before and after exposure trials
  Interventions: Behavioral: reward-focused intervention; Behavioral: exposure; Behavioral: Psychoeducation
- Cognitive flexibility intervention + exposure (Active Comparator): Psychoeducation Cognitive Flexibility based on Unified Protocol of emotional disorders Exposure & cognitive flexibility interventions before and after exposure trials
  Interventions: Behavioral: cognitive flexibility intervention; Behavioral: exposure; Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: reward-focused intervention — Participants complete three interventions based on the Positive Affect Treatment:
  * Finding the silver lining includes attending to and appreciating positive aspects of past events
  * Taking ownership includes identifying the personal behavioral contribution to rewarding past experiences
  * Imagining the positive includes training the prospective, positive imagination of future events
  Participants are asked to practice these interventions at least three times a week (approx. 15 mins each) until the next training session.
  Arms: reward-focused intervention + exposure
Behavioral: cognitive flexibility intervention — This training aims to promote cognitive flexibility in the context of public speaking situations. The intervention is based on the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders.
  Participants will be trained to identify and modify non-adaptive thoughts occurring in the context of public speaking situations.
  Arms: Cognitive flexibility intervention + exposure
Behavioral: exposure — All participants undergo an exposure training session lasting approximately 90 minutes, which includes three exposure trial where participants give a speech, each lasting 5 minutes.
  Exposure exercises are enriched with interventions of the respective treatment group (either reward-focused or cognitive flexibility interventions).
Behavioral: Psychoeducation — All participants received information on anxiety, and the maintenance of anxiety as well as a rationale for the exposure session.

SUMMARY:
The present study aims to examine whether the efficacy of an exposure treatment in individuals with public speaking anxiety can be enhanced by implementing interventions that target reward processes. Optimized exposure enriched with reward-focused interventions will be compared to exposure in combination with interventions targeting cognitive flexibility. The efficacy of the exposure training will be assessed by behavioural and self-report measures of public-speaking anxiety at baseline (before intervention), intermediate-assessment (7-9 days after baseline assessment) and post-assessment (at least 7-9 days after intermediate-assessment). The investigators expect that exposure optimized by implementing reward-focused interventions is more effective in reducing public speaking anxiety compared to exposure in combination with interventions targeting cognitive flexibility.

DETAILED DESCRIPTION:
The present study aims to investigate the efficacy of an optimized exposure training enriched with reward-focused interventions compared to exposure in combination with interventions targeting cognitive flexibility in individuals with elevated public speaking anxiety. Cognitive behavioral therapy offers effective methods for the treatment of various anxiety disorders. However, a substantial number of patients does not benefit from such treatments or experience a return of fear following successful treatment. Emerging evidence underscores the critical involvement of reward processes in fear extinction. Incorporating reward processes in exposure treatments might help to maximize treatment outcomes. In the present study, the investigators will apply reward-focused strategies prior to and during exposure. Strategies are selected to target the core reward processes (i.e., reward anticipation, attainment and learning). Interventions involve finding the silver lining, taking ownership and imagining the positive. Finding the silver lining mainly targets reward attainment (liking) by attending to and appreciating positive aspects of past events. Taking ownership targets liking and reward learning by identifying the personal behavioral contribution to rewarding past experiences. The intervention imagining the positive targets the anticipation of reward (wanting) by training the prospective, positive imagination of future events. The investigators will use an active control group, in which a training of cognitive flexibility (CF; Barlow et al., 2018) will be performed. This training aims to promote cognitive flexibility in the context of public speaking situations. Participants will be trained to identify and modify non-adaptive thoughts (e.g. catastrophizing thoughts). All participants first receive psychoeducation (information on public speaking anxiety, maintenance of anxiety, rationale of exposure training), followed by either reward-focused interventions (Finding the Silver Lining, Taking Ownership, Imagining the Positive) or the CF intervention. Following this session, participants will be asked to practice these interventions between sessions. After one week, exposure in combination with either reward-focused or cognitive flexibility strategies will be performed. Symptom improvement will be assessed at the baseline assessment (i.e., before interventions), at the intermediate-assessment (i.e., before the exposure sessions) and at post assessment (i.e., one week after the exposure sessions). The aim of this randomized controlled trial in individuals with elevated public speaking anxiety is to investigate whether the exposure combined with reward-focused interventions is more effective in reducing public speaking anxiety compared to extinction training combined with cognitive flexibility training.

ELIGIBILITY:
Inclusion Criteria:

* Proficient in the German language.
* Elevated levels of anxiety and avoidance of public speaking situations as indicated by a score of > 5 and > 4, respectively, on a scale from 0 to 8 using the following items:

How anxious would you feel giving a formal speech before a live audience? How likely would you be to avoid taking a class that required taking an oral presentation?

Exclusion Criteria:

* severe cardiovascular, respiratory or neurological diseases
* current psychotherapeutic/psychiatric treatment
* Intention to start psychotherapeutic/psychiatric treatment
* current suicidal ideations
* psychotic symptoms (lifetime)
* current psychopharmacological medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Personal Report of Public Speaking Anxiety (PRPSA) | Change from baseline to intermediate-assessment (i.e., 7-9 days later) to post assessment (i.e., at least 7 days after intermediate-assessment)
  34-item scale for measuring fear of public speaking, each item is rated on a 5-item Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Cronbach's alpha has been shown to range from 0.84 to 0.97. High scores on the scale reflect higher fear of public speaking
Behavioral Approach Test (BAT) | Change from baseline to intermediate-assessment (i.e., 7-9 days later) to post assessment (i.e., at least 7 days after intermediate-assessment)
  Rated fear on a scale from 0 (no fear) to 100 (severe fear) during oral presentation.

SECONDARY OUTCOMES:
Temporal Experience of Pleasure Scale (TEPS) | Change from baseline to intermediate-assessment (i.e., 7-9 days later) to post assessment (i.e., at least 7 days after intermediate-assessment)
  the scale measures individual trait dispositions in anticipatory and consummatory experiences of pleasure, it consists of a 10-item anticipatory pleasure scale and an 8-item consummatory pleasure scale, response format is a 6-point Likert scale from 1 (very false for me) to 6 (very true for me).
Positive and Negative Affect Schedule (PANAS) | Change from baseline to intermediate-assessment (i.e., 7-9 days later) to post assessment (i.e., at least 7 days after intermediate-assessment)
  )]: The PANAS consists of two 10-items scales, one measuring Positive Affect (PA) and the other measuring Negative Affect (NA). Each item on the measure is rated on a 5-point scale (1=not at all; 2=a little; 3=moderately; 4= quite a bit; and 5=extremely). Positive Affect (PA) "reflects the extent to which a person feels enthusiastic, active, and alert". Negative Affect (NA) is a "general dimension of subjective distress and unpleasurable engagement that subsumes a variety of aversive mood states". Higher scores on the PA dimension indicate a greater extent of positive affect, higher scores on the NA dimension indicate a greater extent of negative affect.
Social Phobia Scale (SPS) | Change from baseline to intermediate-assessment (i.e., 7-9 days later) to post assessment (i.e., at least 7 days after intermediate-assessment)
  The SPS "assesses fears of being scrutinised during routine activities", it consists of 20 items with a 5-point Likert scale from 0 (not at all characteristic or true of me) to 4 (extremely characteristic or true of me), higher scores indicating greater distress when undertaking certain activities in the presence of others.
Brief fear of negative evaluations (BFNE-R) | Change from baseline to intermediate-assessment (i.e., 7-9 days later) to post assessment (i.e., at least 7 days after intermediate-assessment)
  the scale is used for measuring fears of negative evaluations. It consists of 12 items with a 5-point Likert scale from 0 (not at all characteristic of me) to 4 (extremely characteristic of me), higher scores indicate a greater fear of negative evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Benke, PhD, Principal Investigator — Philipps University Marburg; Anton Regorius, PhD, Principal Investigator — Philipps University Marburg
Locations (1):
- Philipps-University Marburg, Marburg, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Craske MG, Meuret AE, Ritz T, Treanor M, Dour HJ. Treatment for Anhedonia: A Neuroscience Driven Approach. Depress Anxiety. 2016 Oct;33(10):927-938. doi: 10.1002/da.22490. PMID 27699943
- [Background] Craske MG, Meuret AE, Ritz T, Treanor M, Dour H, Rosenfield D. Positive affect treatment for depression and anxiety: A randomized clinical trial for a core feature of anhedonia. J Consult Clin Psychol. 2019 May;87(5):457-471. doi: 10.1037/ccp0000396. PMID 30998048
- [Background] Barlow DH, Farchione TJ, Bullis JR, Gallagher MW, Murray-Latin H, Sauer-Zavala S, Bentley KH, Thompson-Hollands J, Conklin LR, Boswell JF, Ametaj A, Carl JR, Boettcher HT, Cassiello-Robbins C. The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders Compared With Diagnosis-Specific Protocols for Anxiety Disorders: A Randomized Clinical Trial. JAMA Psychiatry. 2017 Sep 1;74(9):875-884. doi: 10.1001/jamapsychiatry.2017.2164. PMID 28768327